CLINICAL TRIAL: NCT04338373
Title: Open Prospective With Historical Control Clinical Study of 0.01 % Atropine Sulfate Effectiveness in Controlling of Myopia Progression in Children
Brief Title: Effectiveness of 0.01% Atropine Sulfate Solution in Controlling of Myopia Progression in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The V.P. Vyhodcev Eye Hospital (Other)
Responsible Party: Principal Investigator, Daria Afanasyeva, Principal Investigator, The V.P. Vyhodcev Eye Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01
Record Dates: First submitted 2020-04-04; First posted 2020-04-08 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Myopia
Keywords: myopia; low dose atropine; progressive myopia; atropine in non-asian population
MeSH Terms: conditions — Myopia; Myopia, Degenerative

STUDY DESIGN:
Intervention Model Description: Open prospective clinical trial with historical control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental): 0.01% Atropine Sulfate solution in "Comfort Drops", nightly instillations to both eyes
  Interventions: Combination Product: 0.01% Atropine sulfate solution in "Comfort Drops" ("AVIZOR S.A.", Spain)

INTERVENTIONS:
Combination Product: 0.01% Atropine sulfate solution in "Comfort Drops" ("AVIZOR S.A.", Spain) — nightly instillations of 0.01% Atropine sulfate solution in "Comfort Drops" ("AVIZOR S.A.", Spain) in both eyes for 12 months

SUMMARY:
Increasing number of myopic children and significant complications of high myopia enhance the necessity of effective control strategy. Instillations of low-dose atropine have been shown to reduce myopia progression in Asian populations but its effect in non-Asian populations is still unclear. This open prospective study with historical control is designed to investigate if 0.01% atropine can reduce myopia progression in Russian children, taking into account a change of difference between manifest and cycloplegic refraction, as well as, myopia progression rate at the time of recruitment.

DETAILED DESCRIPTION:
The study is designed to test the following hypotheses:

* 0.01% atropine one drop nightly is safe and with no significant side effects.
* nightly instillations of 0.01% atropine does not influence tear production.
* 0.01% atropine one drop nightly reduces the progression of childhood myopia in Russian children.
* nightly instillations of 0.01% atropine decreases the manifest refraction and, consequently, difference between manifest and cycloplegic refractions.
* effectiveness of 0.01% atropine depends on the age and myopia progression rate at the time the therapy was started.

ELIGIBILITY:
Inclusion Criteria:

* myopia progression rate of 0.5D or more per year;
* myopia with astigmatism of 1.0D or less;
* axial length and cycloplegic refraction data obtained 6 months before recruiting or earlier
* signed informed consent.

Exclusion Criteria:

* congenital myopia;
* onset of myopia at 6 years old or earlier;
* allergic reactions to any eye drops in anamnesis;
* concomitant eye disorders, including strabismus.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
change in axial length | baseline - 12 months
  Change in axial length elongation from baseline to 12 months, as measured using IOLMaster, compared with historical data
change in myopic progression rate | baseline - 12 months
  Change in myopic progression rate measured as the difference between cycloplegic refraction from baseline to 12 months, compared with historical data.

SECONDARY OUTCOMES:
change in difference between manifest and cycloplegic refractions | baseline - 12 months
  change in difference between manifest and cycloplegic (tropicamide 0.5%) refractions, measured with autorefractometer, compared with historical data
change in positive relative accommodation | baseline - 12 months
  change in positive relative accommodation, measured in maximal spectacles correction by using concave lenses until the image blurs
tear production | baseline - 12 months
  result of Schirmer I test

CONTACTS AND LOCATIONS:
Locations (1):
- The V.P. Vyhodcev Eye Hospital, Omsk, Russia

IPD SHARING:
Plan to Share IPD: No